CLINICAL TRIAL: NCT04602767
Title: Low Dose Vasopressin vs Phenylephrine in Cardiac Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Jordan Goldhammer, Associate Professor of Anesthesiology, Thomas Jefferson University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20D.847
Record Dates: First submitted 2020-10-20; First posted 2020-10-26 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Vasopressins; Phenylephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vasopressin (Experimental): Low dose vasopressin as first line vasopressor in cardiac surgery.
  Interventions: Drug: Vasopressin
- Phenylephrine (Experimental): Low dose phenylephrine as first line vasopressor in cardiac surgery
  Interventions: Drug: Phenylephrine

INTERVENTIONS:
Drug: Vasopressin — Vasopressin titrated 0.01 U/min up to 0.04 U/min for MAP < 65 mmHg
  Other Names: Pitressin
  Arms: Vasopressin
Drug: Phenylephrine — Phenylephrine titrated 0.25 mcg/kg/min up to 1.0 mcg/kg/min for MAP < 65 mmHg
  Other Names: Neosynephrine
  Arms: Phenylephrine

SUMMARY:
This is a randomized, open label study to investigate vasopressin versus phenylephrine as a first line pressor in cardiac surgery. All patients >18 years of age presenting for coronary artery bypass graft (CABG), valve surgery, or combined CABG and valve surgery will be screened for inclusion. Patients with ejection fraction < 35%, > moderate pulmonary hypertension, > mild right ventricular dysfunction, a planned radial arterial graft, or circulatory arrest will be excluded. Patients will be randomized to receive either vasopressin or phenylephrine as the first line vasopressor during the perioperative period to maintain mean arterial blood pressure >65 mmhg. Primary outcome is acute kidney injury. Secondary outcomes are 30-day mortality, stroke, myocardial infarction, re-operation, sternal infection, atrial fibrillation, intensive care unit length of stay, and total vasopressor hours.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Coronary artery bypass graft (CABG), valve, or combined CABG and valve surgery

Exclusion Criteria:

* Ejection fraction < 35%
* > moderate pulmonary hypertension
* > mild right ventricular dysfunction
* Radial arterial graft
* Circulatory arrest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-10-15 (Actual); Primary Completion 2024-05-29 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with acute kidney injury | 5 Days
  KDIGO criteria

SECONDARY OUTCOMES:
Number of patients with 30-Day Mortality | 30 Days
  Number of patients with 30-Day Mortality
Number of patients with reoperation | 5 Days
  Number of patients with reoperation
Number of patients with sternal Infection | 5 Days
  Number of patients with sternal Infection
Number of patients with Atrial Fibrilation | 5 Days
  Number of patients with Atrial Fibrilation
ICU Length of Stay | 5 Days
  Total ICU Length of Stay
Total Vasopressor Hours | 5 Days
  Total Vasopressor Hours

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson Univesity, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No